CLINICAL TRIAL: NCT02499315
Title: A Randomized, Double-blind, Placebo-controlled, Ascending Multiple-dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AMG 357 in Female Subjects With Rheumatoid Arthritis
Brief Title: Study to Evaluate the Safety, Tolerability, and Action of AMG 357 in Females With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study has stopped due to a decision by Amgen to terminate the program
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20110247
Record Dates: First submitted 2015-04-10; First posted 2015-07-16 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 357 (Experimental)
  Interventions: Drug: AMG 357
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 357 — Oral tablets in 20 count bottles. Dose strengths include 5, 25, and 50 mg tablets.
  Arms: AMG 357
Drug: Placebo — Oral tablets in 20 count bottles. Dose strengths include 5, 25, and 50 mg tablets.
  Arms: Placebo

SUMMARY:
The purpose of the study is to find out if AMG 357 is safe and tolerated by women with Rhematoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subject provided informed consent.
* Rheumatoid arthritis present for ≥ 3 months.
* Global functional class I, II, or III.
* History of or positive for, Rheumatoid Arthritis
* Taking methotrexate consecutively for ≥ 12 weeks and on a stable dose at 10-25 mg weekly.
* Subjects currently taking NSAIDs or oral corticosteroids.
* Normal ECG values
* Immunizations up to date.

Exclusion Criteria:

* Positive Hepatitis B, Hepatitis C, Positive HIV
* Sensitivity to any of the products or components to be administered.
* Malignancy within 3 years
* Presence of recurrent or chronic infections
* Evidence of infections within the 30 days prior to randomization
* Presence of a serious infection
* Prosthetic joint infection within 3 years or native joint infection within 1 year
* History of exposure to tuberculosis without a history of prophylactic treatment
* Class IV RA.
* Felty's syndrome
* Chronic pelvic pain or hemorrhagic ovarian cyst within 3 years
* Any bleeding disorder that is clinically significant
* Low white blood cell or neutrophil count
* Elevated serum creatinine clearance
* Low hemoglobin and platelet count
* Received live vaccines within 3 months of first dose
* Alcohol and/or substance abuse within past 12 months
* Blood donation within 60 days
* Positive urine screen for drugs of abuse
* Any prior use of rituximab in the last 6 months (or other B cell depleting agents) and CD19 levels < lower limits of normal
* Use of a weekly or bimonthly biologic within 2 weeks or monthly biologic agents within 4 weeks
* Corticosteroid injections for acute RA flare within 4 weeks
* Grapefruit juice or grapefruit containing products within 7 days of first dose.
* All herbal medicines, vitamins, and supplements within the 30 days
* The use of any experimental/investigational biologic DMARD unless off agent for 3 months; or off for 6 months for B cell depleting agents
* Known GI disease or GI procedures
* Women of reproductive potential who are unwilling to practice birth control
* Women who are pregnant/lactating/breastfeeding
* Subject with IgG levels < lower limit of normal at screening

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The number of subjects reporting of treatment-emergent adverse events or clinically significant changes in physical examinations, vital signs, laboratory safety tests, and ECGs | 1 year

SECONDARY OUTCOMES:
AMG 357 pharmacokinetic profile (eg, plasma concentration, maximum observed concentration [Cmax], time at Cmax [Tmax], and area under the concentration-time curve [AUC]) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Dallas, Texas

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com